CLINICAL TRIAL: NCT06814782
Title: Effects of Action Observation Training and Motor Imagery Delivered by Telerehabilitation on Mobility, Posture and Brain Plasticity in Patients with Parkinson's Disease
Brief Title: Effects of Action Observation Training and Motor Imagery Delivered by Telerehabilitation in Patients with Parkinson's Disease
Acronym: TeleAOTPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF24/01; PRIN: 2022FABKJ5_2 (Other Grant/Funding Number: PNRR - Next Generation EU)
Record Dates: First submitted 2025-01-10; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Action Observation; Motor Imagery; Telerehabilitation; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Action Observation Training Group (AOT) (Experimental): Patients in this group will be exposed to four video presentations showing movements with different degrees of focal vs. postural components. The patients will imitate immediately after watching.
  Interventions: Other: Action Observation Training
- Action Observation and Motor Imagery Group (AOMI) (Experimental): Patients in this group will be exposed to four video presentations showing movements with different degrees of focal vs. postural components. The patients will mentally rehearse what they saw in the videos immediately after watching.
  Interventions: Other: Action Observation and Motor Imagery
- Control group (Active Comparator): Patients in this group will be exposed to four video presentations showing landscape. Patients will perform the same exercise of AOT groupimmediately after watching.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Action Observation Training — Action Observation Training (AOT) consists of patients observing videos of specific movements, followed by practice of those movements
  Other Names: AOT; Action Observation Therapy
  Arms: Action Observation Training Group (AOT)
Other: Action Observation and Motor Imagery — Action Observation and Motor Imagery (AOMI) consists of patients observing videos of specific movements, followed by mental rehearsal of those movements
  Other Names: AOMI
  Arms: Action Observation and Motor Imagery Group (AOMI)
Other: Exercise — After watching a landscape video, patients will have to perform specific postural and balance exercises
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy on motor and postural tasks of Action Observation Training (AOT) and Action Observation combined with Motor Imagery (AOMI) delivered by telerehabilitation in patients with Parkinson Disease.

* The primary endpoint will be mobility measured with the Timed Up and Go (TUG) test (differences before and after telerehabilitation treatment period).
* In addition, clinical and functional measures, instrumental analysis of gait and posture, and Magnetic Resonance Imaging (MRI) correlates will be assessed.

Participants will be asked to undergo 24 telerehabilitation sessions, cadenced 3 per week, over an 8-week period. In the two experimental groups (AOT and AOMI), each telerehabilitation session will encompass 4 motor tasks, each containing the observation of a video clip immediately followed by the patient's execution or imagination of the same exercises. Patients in the control group will be instructed to perform the same exercises after watching videos showing landscapes

DETAILED DESCRIPTION:
The project is a a single center randomised controlled trial and aims to investigate the efficacy of Action Observation Training (AOT) and Action Observation with Motor Imagery (AOMI) delivered via telerehabilitation for improving motor and postural functions in patients with Parkinson's Disease (PD). Additionally, the study seeks to explore the cortical plasticity induced by AOMI using neuroimaging techniques. The primary outcome measure will be the Timed Up and Go (TUG) test, evaluating changes in mobility before and after the 8-week telerehabilitation intervention. Secondary outcomes include clinical and functional assessments, gait and gait initiation analysis and posture analysis. For gait and gait initiation analysis and posture analysis a sex and age matched healthy subjects cohort will be included. It will be also assessed postural motor resonance in AOT group and control group during action observation at all time point and results compared to sex and age match healthy cohort. Finally last 15 recruited patients of AOMI and control group will undergo fMRI investigation.

The study will enroll 60 PD patients, each meeting specific criteria. Participants will be randomly assigned to one of three groups: 1) AOT, 2) AOMI, or 3) a control group. The intervention will consist of 24 telerehabilitation sessions over 8 weeks (3 sessions per week). Each AOT and AOMI session will include four motor tasks, where patients will watch 3-minute video clips, followed by either performing (AOT) or imagining (AOMI) the exercise for 1 minute. Each task will be repeated twice, resulting in a 32-minute session. Exercises will focus on gait and balance, commonly used in PD rehabilitation. The control group will perform similar exercises after watching videos of neutral content, such as landscapes.

Assessments will be conducted by blinded evaluators at three time points: baseline (T0), immediately after the intervention period (T8W), and three months post-intervention (T5M).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of clinically definite PD according to the Movement Disorders Society criteria
* Hoehn and Yahr scale <4
* Montreal Cognitive Assessment, MoCA ≥ 26
* a stable medication regimen for at least 4 weeks.

Exclusion Criteria:

* Systemic, psychiatric, or other neurological illnesses influencing motor or functional performance
* a history of substance abuse influencing cognition or compliance
* visual disturbances
* head tremor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go test | From enrollment to the end of treatment at 8 weeks
  Patients will be instructed to stand up from a chair, walk 3 meters, turn, and return to sit down. The time taken to complete the task will be recorded.

SECONDARY OUTCOMES:
Timed Up and Go test | From enrollment to the end of follow-up at 3 months after end of training
  Patients will be instructed to stand up from a chair, walk 3 meters, turn, and return to sit down. The time taken to complete the task will be recorded.
Timed Up and Go test | From end of training to the end of follow-up at 3 months after end of training
  Patients will be instructed to stand up from a chair, walk 3 meters, turn, and return to sit down. The time taken to complete the task will be recorded.
Movement Disorders Society Unified PD Rating Scale | From enrollment to the end of treatment at 8 weeks
  It's a scale that invenstigates behavioural, motor and functional status of PD patients. The scale is divided in 4 parts and higher score represents worsebehavioural, motor and functional status.
Movement Disorders Society Unified PD Rating Scale | From enrollment to the end follow-up (3 months after end of training)
  It's a scale that invenstigates behavioural, motor and functional status of PD patients. The scale is divided in 4 parts and higher score represents worsebehavioural, motor and functional status.
Movement Disorders Society Unified PD Rating Scale | From end of training to the end follow-up (3 months after end of training)
  It's a scale that invenstigates behavioural, motor and functional status of PD patients. The scale is divided in 4 parts and higher score represents worsebehavioural, motor and functional status.
Functional Independence Measure (FIM) | From enrollment to the end of treatment at 8 weeks
  Functional Independence Measure quantifies autonomy during daily activities
Functional Independence Measure (FIM) | From enrollment to the end follow-up (3 months after end of training)
  Functional Independence Measure quantifies autonomy during daily activities
Functional Independence Measure (FIM) | From end of treatment to the end of follow-up (3 months after end of treatment)
  Functional Independence Measure quantifies autonomy during daily activities
Parkinson's disease Questionnaire - 39 items (PDQ-39) | From enrollment to the end of treatment at 8 weeks
  Parkinson's disease Questionnaire - 39 items (PDQ-39) investigates quality of life in PD patients.
Parkinson's disease Questionnaire - 39 items (PDQ-39) | From enrollment to the end follow-up (3 months after end of treatment)
  Parkinson's disease Questionnaire - 39 items (PDQ-39) investigates quality of life in PD patients.
Parkinson's disease Questionnaire - 39 items (PDQ-39) | From end of treatment to the end of follow-up (3 months after end of treatment)
  Parkinson's disease Questionnaire - 39 items (PDQ-39) investigates quality of life in PD patients.
Mini-BEST Test | From enrollment to the end of treatment at 8 weeks
  Mini-BEST Test investigates dynamic balance control.
Mini-BEST Test | From enrollment to the end follow-up (3 months after end of treatment)
  Mini-BEST Test investigates dynamic balance control.
Mini-BEST Test | From end of treatment to the end of follow-up (3 months after end of treatment)
  Mini-BEST Test investigates dynamic balance control.
10-Meter Walking test | From enrollment to the end of treatment at 8 weeks
  10-Meter Walking test investigates spontaneous and maximum walking speed.
10-Meter Walking test | From enrollment to the end follow-up (3 months after end of treatment)
  10-Meter Walking test investigates spontaneous and maximum walking speed.
10-Meter Walking test | From end of treatment to the end of follow-up (3 months after end of treatment)
  10-Meter Walking test investigates spontaneous and maximum walking speed.
6-Minute Walking test | From enrollment to the end of treatment at 8 weeks
  6-Minute Walking test investigates walking endurance.
6-Minute Walking test | From enrollment to the end follow-up (3 months after end of treatment)
  6-Minute Walking test investigates walking endurance.
6-Minute Walking test | From end of treatment to the end of follow-up (3 months after end of treatment)
  6-Minute Walking test investigates walking endurance.
Freezing of Gait Questionnaire | From enrollment to the end of treatment at 8 weeks
  Freezing of Gait Questionnaire investigates freezing of gait episodes during daily life
Freezing of Gait Questionnaire | From enrollment to the end follow-up (3 months after end of treatment)
  Freezing of Gait Questionnaire investigates freezing of gait episodes during daily life
Freezing of Gait Questionnaire | From end of treatment to the end follow-up (3 months after end of treatment)
  Freezing of Gait Questionnaire investigates freezing of gait episodes during daily life

OTHER OUTCOMES:
Gait and gait initiation analysis | From enrollment to the end of treatment at 8 weeks
  Gait and gait initiation analysis measure the kinematic parameters of gait and the Anticipatory Postural Adjustments
Gait and gait initiation analysis | From enrollment to the end follow-up (3 months after end of treatment)
  Gait and gait initiation analysis measure the kinematic parameters of gait and the Anticipatory Postural Adjustments
Posture analysis | From enrollment to the end of treatment at 8 weeks
  Change of postural motor resonance of the mirror neuron system during Action Observation through H-reflex assessment
Posture analysis | From enrollment to the end follow-up (3 months after end of treatment)
  Change of postural motor resonance of the mirror neuron system during Action Observation through H-reflex assessment
Functional Magnetic Resonance Imaging | From enrollment to the end of treatment at 8 weeks
  fMRI investigates brain plasticity and functional reorganization

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided